CLINICAL TRIAL: NCT01969955
Title: A Phase II Trial of Nab-paclitaxel as Second-line Therapy in Locally Advanced or Metastatic Squamous Lung Cancer After Failure of Platinum Doublet (Except Pemetrexed) Therapy
Brief Title: Nab-paclitaxel as Second-line Therapy in Locally Advanced or Metastatic Squamous Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LI Junling, Professor and chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-031
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Squamous Cell Carcinoma of Lung
Keywords: nanoparticle albumin-bound paclitaxel; Squamous Cell Carcinoma of Lung
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nanoparticle albumin-bound paclitaxel (Experimental): Nanoparticle albumin-bound paclitaxel is given at 130 mg/m2 intravenously on day 1 and 8, every 21 days.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — Nanoparticle albumin-bound paclitaxel is given at 130 mg/m2 intravenously on day 1 and 8, every 21 days.
  Other Names: Abraxane, nab-paclitaxel

SUMMARY:
The purpose of this study is to determine the efficacy of nab-paclitaxel monotherapy in previously treated advanced or metastatic squamous lung cancer.

DETAILED DESCRIPTION:
Nanoparticle albumin-bound paclitaxel (nab-paclitaxel) is a novel, solvent-free, albumin-bound nanoparticle form of paclitaxel designed to avoid problems associated with solvents used in Taxol. And albumin-bound paclitaxel was characterized with high tolerated doses with greater efficacy, and with greater concentration in tumor tissue compared with normal tissues. A multicenter randomized controled trial (coded as CA031) showed that nab-paclitaxel in combination with carboplatin had higher response rate than traditional paclitaxel plus carboplatin, especially in squamous lung cancer. This is a single center, non-randomized, open-label Phase II clinical study to investigate the efficacy and tolerability of nab-paclitaxel monotherapy in previously treated advanced or metastatic squamous lung cancer after failure of platinum-based doublet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form;
2. Age no less than 18 years;
3. Histologically confirmed locally advanced or metastatic squamous lung cancer;
4. Eastern Cooperative Oncology Group (ECOG) 0-2 with life expectation of no less than 12 weeks;
5. RECIST measurable lesions;
6. Disease progression after failure of platinum-based doublet therapy;
7. Adequate liver/renal/bone marrow function;
8. Human Chorionic Gonadotropin (HCG) test negative for female with contraception measures until 3 months after study end;
9. Compliance, and can be followed up regularly.

Exclusion Criteria:

1. Pregnant or breast-feeding female, or not willing to take contraception measures during study;
2. Radiotherapy within 30 days, systematic therapy within 21 days;
3. Serious infection requiring antibiotics intervention during recruitment;
4. Allergic to study drug;
5. Require concurrent biological target therapy;
6. More than grade 1 neuropathy;
7. Uncontrolled brain metastasis or mental illness;
8. Congestive heart failure, uncontrolled cardiac arrhythmia, etc;
9. Other malignancy within 5 years;
10. Can't be followed up or obey protocol;
11. Ineligible by the judge of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to one year
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).

SECONDARY OUTCOMES:
progression-free survival | up to 15 months
  Measure of time from study treatment to disease progression or death.
Overall survival | up to 2 years
  Measure of time from study treatment to patient's death or lost to follow-up.
Quality of life | up to 15 months
  Determine the score change of quality of life between pre- and post-treatment.
Safety and tolerability | up to 18 months
  Percentage of patients who experience an adverse event during this study.

OTHER OUTCOMES:
secreted protein acidic and rich in cysteine (SPARC) expression level in tumor issues | up to 15 months
  Correlationship between secreted protein acidic and rich in cysteine (SPARC) expression in tumor issue and the efficacy of nab-paclitaxel or prognosis of patients

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer institute and hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China